CLINICAL TRIAL: NCT04612049
Title: Immersive Virtual Reality for Visuo-motor Integration Skill Assessment in Children With Hemiplegia
Brief Title: Immersive Virtual Reality for Visuo-motor Integration Skill Assessment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator changed sites
Sponsor: Northeastern University (Other)
Collaborators: MaineHealth (Other); Massachusetts General Hospital (Other); Spaulding Rehabilitation Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 412575-19357; P2CHD101912 (NIH)
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Cerebral Palsy; Hemiplegia
Keywords: Virtual Reality; Visual-Motor Integration; Feasibility
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with hemiplegia (Experimental): 40 children with hemiplegia, 7-16 years-old at Gross Motor Function Classification System (GMFCS) Levels I-III and Manual Ability Classification System (MACS) Levels I-II will be recruited as participants. This age range was chosen based on our preliminary research in which children under the age of 7 had difficulty attending to repetitive task practice. Individuals will be recruited without regard to race or ethnicity. Our goal is to have a study sample that is 50% male and 50% female, and approximates the population of the Greater Boston, MA region.
  Interventions: Device: Immersive virtual reality visuo-motor skill assessment
- Typically developing children (Experimental): 40 typically developing children, 7-16 years-old.
  Interventions: Device: Immersive virtual reality visuo-motor skill assessment

INTERVENTIONS:
Device: Immersive virtual reality visuo-motor skill assessment — Visuo-motor skill assessment in an immersive 3D virtual environment using a head-mounted display.

SUMMARY:
A significant deficit affecting nearly half of children with hemiplegia is visual-motor integration, or eye-hand coordination. Children have difficulties integrating visual and motor information to effectively plan and execute movements. Visual-motor impairments are detrimental because they affect accuracy of reaching and grasping, which are movements involved in feeding, writing, and sports participation, among many other daily life activities. Although paper-and-pencil and touchscreen computer assessments exist, these fail to evaluate impairments under realistic, 3D conditions. This assessment barrier leads to significant gaps in knowledge the influence of these impairments on children's performance of functional activities.

We will use immersive virtual reality (VR) delivered using a head-mounted display (HMD) to address this gap. Because it is fully visually immersive, VR makes interactions similar to real world performance. These features enable HMD-VR to offer more natural assessment conditions. HMD-VR may help us gain important new knowledge about functional movement deficits in children with hemiplegia.

The purpose of this study is to evaluate low-cost HMD-VR as a realistic assessment tool for visual-motor integration deficits in children with hemiplegia. The long-term goals of our research program are to: 1) Inform clinical decision-making practices by providing families and clinicians with precise, accurate information about children's abilities; and 2) Generate new knowledge about visual-motor integration impairments to enhance the effectiveness of both virtual and conventional rehabilitation interventions. We will recruit 40 children with hemiplegia aged 7-16 years at GMFCS Levels I-III and Manual Ability Classification System levels I-II for testing sessions of seated paper-and-pencil, touchscreen computer and HMD-VR visual-motor integration tasks at 3 clinical sites We will measure feasibility using counts of enrollment, side-effects and protocol completion. Visual-motor integration is quantified in the paper-and-pencil task via standardized score and in touchscreen and HMD-VR tasks using equivalent temporal and spatial eye and hand metrics. This pilot study will generate descriptive estimates of differences in visual-motor performance under conditions of differing 3D realism. This work is the first step towards the ultimate goal of a valid assessment method informing new VR-based treatment options for children with hemiplegia.

DETAILED DESCRIPTION:
In a private testing room at the testing site, children will complete descriptive functional sensory-motor tests with a registered physical therapist. They will then complete the paper-and-pencil visual-motor integration test (Beery-Buktenica Test of Visual Motor Integration) while seated comfortably. They will then undertake the visuomotor integration tasks using a touch screen computer, completing 5 trials of each of 3 target positions under visual-only, motor-only, and visual-motor integration conditions. The task will be displayed on a 20" HP Spectre touch-screen laptop with an RTX 960 graphics card. Eye-tracking will be undertaken using a Tobii Nano which integrates with Unity software. Kinematics of hand movement during reach to touch as well as head movements will be collected using an Orbbec Astra depth-sensing camera. Accuracy of touch is recorded by custom-written software tracking X-Y touch coordinates on the screen. All data collection modalities are synced and integrated using LabVIEW.

Children will then complete the same tasks in the 3D HMD virtual environment. We will use the VIVE Pro EYE, the leading commercially-available immersive VR system, which has with a 110 degree trackable field of view and an embedded eye tracker. Arm movements are tracked by lightweight trackers attached via Velcro arm band to children's forearms and ManusVR motion tracking gloves worn on the hands. Head movements are tracked by position sensors in the HMD. Trackers and gloves enable upper extremity interaction with objects in the virtual world. An Alienware m15 gaming laptop with an NVIDA GeForce RTX 2060 graphics card will run the task. Following the visual-only, motor-only, and visual-motor integration tasks, children will complete a new visual-motor integration task involving virtual object transport, where they will grasp a virtual object and transport it to a new location in the virtual environment. Finally, they will complete the object transport task in a more audiovisually-complex virtual environment in the HMD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemiplegia (due to CP or stroke)
* Gross Motor Function Classification System (GMFCS) Levels I-III
* Manual Ability Classification System (MACS) Levels I-II
* Ability to read and write English.
* Sufficient hearing, vision and cognition to respond to auditory and visual cues.

Exclusion Criteria:

* Greater than 10-degree elbow or shoulder flexion contracture in the affected arm
* Uncorrected visual deficits (e.g., homonymous hemianopsia, oculomotor disturbance, or cortical visual impairment)
* Uncontrolled photosensitive seizures (occurrence of at least one seizure in the last 3 months)
* Hemineglect
* Cognitive impairments that would prohibit participation (as judged by a parent)

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Levac, PhD, Principal Investigator — Northeastern University
Locations (3):
- United States (3):
  - Maine Health, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Spaulding Rehabilitation, Salem, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ronnqvist L, Rosblad B. Kinematic analysis of unimanual reaching and grasping movements in children with hemiplegic cerebral palsy. Clin Biomech (Bristol). 2007 Feb;22(2):165-75. doi: 10.1016/j.clinbiomech.2006.09.004. Epub 2006 Oct 27. PMID 17070630
- [Background] Mackey AH, Walt SE, Stott NS. Deficits in upper-limb task performance in children with hemiplegic cerebral palsy as defined by 3-dimensional kinematics. Arch Phys Med Rehabil. 2006 Feb;87(2):207-15. doi: 10.1016/j.apmr.2005.10.023. PMID 16442974
- [Background] Graham HK, Rosenbaum P, Paneth N, Dan B, Lin JP, Damiano DL, Becher JG, Gaebler-Spira D, Colver A, Reddihough DS, Crompton KE, Lieber RL. Cerebral palsy. Nat Rev Dis Primers. 2016 Jan 7;2:15082. doi: 10.1038/nrdp.2015.82. PMID 27188686
- [Background] Shevell MI, Dagenais L, Hall N; REPACQ CONSORTIUM*. The relationship of cerebral palsy subtype and functional motor impairment: a population-based study. Dev Med Child Neurol. 2009 Nov;51(11):872-7. doi: 10.1111/j.1469-8749.2009.03269.x. Epub 2009 Mar 11. PMID 19416339
- [Background] Ego A, Lidzba K, Brovedani P, Belmonti V, Gonzalez-Monge S, Boudia B, Ritz A, Cans C. Visual-perceptual impairment in children with cerebral palsy: a systematic review. Dev Med Child Neurol. 2015 Apr;57 Suppl 2:46-51. doi: 10.1111/dmcn.12687. PMID 25690117
- [Background] James S, Ziviani J, Ware RS, Boyd RN. Relationships between activities of daily living, upper limb function, and visual perception in children and adolescents with unilateral cerebral palsy. Dev Med Child Neurol. 2015 Sep;57(9):852-7. doi: 10.1111/dmcn.12715. Epub 2015 Feb 23. PMID 25703777
- [Background] Mallory K, Barton K, Woodhouse J, Bernstein J, Greenspoon D, Reed N. Occupational Performance Issues of Children with Hemiplegia after Acquired Brain Injury. Phys Occup Ther Pediatr. 2020;40(3):279-293. doi: 10.1080/01942638.2019.1675845. Epub 2019 Oct 14. PMID 31608806
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Oskoui M, Coutinho F, Dykeman J, Jette N, Pringsheim T. An update on the prevalence of cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2013 Jun;55(6):509-19. doi: 10.1111/dmcn.12080. Epub 2013 Jan 24. PMID 23346889
- [Background] Chiu HC, Ada L. Constraint-induced movement therapy improves upper limb activity and participation in hemiplegic cerebral palsy: a systematic review. J Physiother. 2016 Jul;62(3):130-7. doi: 10.1016/j.jphys.2016.05.013. Epub 2016 Jun 17. PMID 27323932
- [Background] Hoare BJ, Wallen MA, Thorley MN, Jackman ML, Carey LM, Imms C. Constraint-induced movement therapy in children with unilateral cerebral palsy. Cochrane Database Syst Rev. 2019 Apr 1;4(4):CD004149. doi: 10.1002/14651858.CD004149.pub3. PMID 30932166
- [Background] Hoare B, Greaves S. Unimanual versus bimanual therapy in children with unilateral cerebral palsy: Same, same, but different. J Pediatr Rehabil Med. 2017;10(1):47-59. doi: 10.3233/PRM-170410. PMID 28339410
- [Background] Krajenbrink H, Crichton A, Steenbergen B, Hoare B. The development of anticipatory action planning in children with unilateral cerebral palsy. Res Dev Disabil. 2019 Feb;85:163-171. doi: 10.1016/j.ridd.2018.12.002. Epub 2018 Dec 14. PMID 30557847
- [Background] Gordon AM. Impaired Voluntary Movement Control and Its Rehabilitation in Cerebral Palsy. Adv Exp Med Biol. 2016;957:291-311. doi: 10.1007/978-3-319-47313-0_16. PMID 28035572
- [Background] Saavedra S, Karve SJ, Woollacott M, van Donkelaar P. Eye hand coordination in children with cerebral palsy. Exp Brain Res. 2009 Jan;192(2):155-65. doi: 10.1007/s00221-008-1549-8. Epub 2008 Oct 2. PMID 18830589
- [Background] Fang Y, Wang J, Zhang Y, Qin J. The Relationship of Motor Coordination, Visual Perception, and Executive Function to the Development of 4-6-Year-Old Chinese Preschoolers' Visual Motor Integration Skills. Biomed Res Int. 2017;2017:6264254. doi: 10.1155/2017/6264254. Epub 2017 Dec 31. PMID 29457030
- [Background] Verrel J, Bekkering H, Steenbergen B. Eye-hand coordination during manual object transport with the affected and less affected hand in adolescents with hemiparetic cerebral palsy. Exp Brain Res. 2008 May;187(1):107-16. doi: 10.1007/s00221-008-1287-y. Epub 2008 Jan 30. PMID 18231781
- [Background] Harvey EM, Leonard-Green TK, Mohan KM, Kulp MT, Davis AL, Miller JM, Twelker JD, Campus I, Dennis LK. Interrater and Test-Retest Reliability of the Beery Visual-Motor Integration in Schoolchildren. Optom Vis Sci. 2017 May;94(5):598-605. doi: 10.1097/OPX.0000000000001068. PMID 28422801
- [Background] Weiss PL, Rand D, Katz N, Kizony R. Video capture virtual reality as a flexible and effective rehabilitation tool. J Neuroeng Rehabil. 2004 Dec 20;1(1):12. doi: 10.1186/1743-0003-1-12. PMID 15679949
- [Background] Levac DE, Huber ME, Sternad D. Learning and transfer of complex motor skills in virtual reality: a perspective review. J Neuroeng Rehabil. 2019 Oct 18;16(1):121. doi: 10.1186/s12984-019-0587-8. PMID 31627755
- [Background] Levac D, Glegg S, Colquhoun H, Miller P, Noubary F. Virtual Reality and Active Videogame-Based Practice, Learning Needs, and Preferences: A Cross-Canada Survey of Physical Therapists and Occupational Therapists. Games Health J. 2017 Aug;6(4):217-228. doi: 10.1089/g4h.2016.0089. PMID 28816511
- [Background] Spodick DH. Accuracy of nongeometric pulsed Doppler cardiac output. Am J Cardiol. 1994 Feb 15;73(5):421. doi: 10.1016/0002-9149(94)90031-0. No abstract available. PMID 8109566
- [Background] Robert MT, Levin MF. Validation of reaching in a virtual environment in typically developing children and children with mild unilateral cerebral palsy. Dev Med Child Neurol. 2018 Apr;60(4):382-390. doi: 10.1111/dmcn.13688. Epub 2018 Feb 10. PMID 29427357
- [Background] de Mello Monteiro CB, Massetti T, da Silva TD, van der Kamp J, de Abreu LC, Leone C, Savelsbergh GJ. Transfer of motor learning from virtual to natural environments in individuals with cerebral palsy. Res Dev Disabil. 2014 Oct;35(10):2430-7. doi: 10.1016/j.ridd.2014.06.006. Epub 2014 Jun 28. PMID 24981192
- [Background] Knaut LA, Subramanian SK, McFadyen BJ, Bourbonnais D, Levin MF. Kinematics of pointing movements made in a virtual versus a physical 3-dimensional environment in healthy and stroke subjects. Arch Phys Med Rehabil. 2009 May;90(5):793-802. doi: 10.1016/j.apmr.2008.10.030. PMID 19406299
- [Background] Subramanian SK, Levin MF. Viewing medium affects arm motor performance in 3D virtual environments. J Neuroeng Rehabil. 2011 Jun 30;8:36. doi: 10.1186/1743-0003-8-36. PMID 21718542
- [Background] Niehorster DC, Li L, Lappe M. The Accuracy and Precision of Position and Orientation Tracking in the HTC Vive Virtual Reality System for Scientific Research. Iperception. 2017 May 18;8(3):2041669517708205. doi: 10.1177/2041669517708205. eCollection 2017 May-Jun. PMID 28567271
- [Background] Fears NE, Bailey BC, Youmans B, Lockman JJ. An Eye-Tracking Method for Directly Assessing Children's Visual-Motor Integration. Phys Ther. 2019 Jun 1;99(6):797-806. doi: 10.1093/ptj/pzz027. PMID 30806663

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Children With Hemiplegia | Typically Developing Children
Started | 12 | 0
Completed | 12 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study timeline due to investigator changing institutions limited collected data with typically developing children.
Groups:
- Total: Total of all reporting groups
Arm/Group | Children With Hemiplegia | Typically Developing Children | Total
Number analyzed (Participants) | 12 | 0 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.25 (2.84) |  | 10.25 (2.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 8
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 12 |  | 12
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 10 |  | 10
  More than one race | 2 |  | 2
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Eye-hand Proximity
Description: Lag between eye end time and hand end time (i.e. eye movement time - hand movement time)
Time Frame: During testing.
Population: Unfortunately our kinematics plan for the 2D task did not enable collection of this outcome measure in the computerized 2D environment and as such we do not report it here for either 2D or immersive 3D.
Arm/Group | Children With Hemiplegia | Typically Developing Children
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Beery-Buktenica VMI Test 6th Edition (Short Form)
Description: The Beery-Bukentica VMI, which is the unabbreviated scale title, is a test of visual-motor integration skills involving geometric design copying tasks. The administration time is 10-15 minutes. Children copy a series of increasingly complex designs using their preferred hand.
  We used the standard score, which ranges from 0 (minimum) to 100 (maximum). Higher scores indicate better VMI skills.
Time Frame: Pre-testing.
Population: No typically developing children were included in the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Children With Hemiplegia | Typically Developing Children
Number analyzed (Participants) | 12 | 0
score on a scale | 83.64 (21.97) |

3. Secondary Outcome: Box and Blocks
Description: he Box and Block Test (BBT) measures unilateral gross manual dexterity. Participants pick up blocks on one side of a wooden box and transport them to the other side, one at a time. The number of blocks successfully transported in one minute is scored. If a block falls or 2 blocks are picked up, it is not counted in the total. The minimum is zero. The maximum number of blocks is 150. A higher number of blocks indicates better gross manual dexterity, otherwise known as fine motor skills.
Time Frame: Pre-testing
Population: No typically developing children took part in the study.
Measure: Mean (Standard Deviation); unit: Number of blocks transported
Arm/Group | Children With Hemiplegia | Typically Developing Children
Number analyzed (Participants) | 12 | 0
Number of blocks transported | 19.75 (16.21) |

ADVERSE EVENTS:
Time Frame: 3 months
Description: No differences
Arm/Group | Children With Hemiplegia | Typically Developing Children
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/0
Other Adverse Events (participants affected / at risk) | 0/12 | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to Investigator changing sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT04612049/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT04612049/ICF_001.pdf